CLINICAL TRIAL: NCT06458803
Title: Efficacy and Safety of Eltrombopag for the Treatment of Refractory Thrombocytopenia Associated With Connective Tissue Disease
Brief Title: Efficacy and Safety of Eltrombopag for Refractory Thrombocytopenia Associated With Connective Tissue Disease
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Lingli Dong, Professor, Tongji Hospital
Other Study IDs: TJ-IRB202404119
Record Dates: First submitted 2024-06-04; First posted 2024-06-14 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Refractory Thrombocytopenia; Connective Tissue Diseases
MeSH Terms: conditions — Thrombocytopenia; Connective Tissue Diseases | interventions — eltrombopag

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- El-treatment: patients receive oral eltrombopag at 25 to 75 mg once daily during the course.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — patients receive oral eltrombopag at 25 to 75 mg once daily according to disease severity，with the treatment of DMARDs at minimal or routine dosages.
  Other Names: Promacta

SUMMARY:
Immune thrombocytopenia (ITP) is a haemorrhagic disorder often associated with CTD. Corticosteroids are the first-line treatment for CTD-associated thrombocytopenia, but not all patients respond well. Eltrombopag is an oral, small molecule thrombopoietin receptor agonist. It interacts with the transmembrane domain of the thrombopoietin receptor and stimulates platelet production. This study is designed to evaluate the efficacy and safety of eltrombopag in patients with refractory CTD-ITP. It is a single-centre, retrospective, observational study involving a cohort of 52 patients diagnosed with CTD-RITP who received eltrombopag between 2013 and 2023. Follow-up data will be systematically collected and analysed to evaluate the therapeutic efficacy and safety of the drug. The study will provide valuable insight into the benefit of eltrombopag in CTD-RITP by reviewing baseline characteristics and performing subsequent clinical assessments to determine drug response and adverse events.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is a hemorrhagic disorder typically attributed to the formation of autoantibodies against platelet antigens. Patients experience decreased platelet count, clinically presenting as purpura, petechiae, mucosal bleeding, and increased menstrual bleeding. ITP is often associated with connective tissue diseases (CTD), with reports indicating a concurrent presence of ITP in 10%-15% of systemic lupus erythematosus (SLE) patients and 7.8% of primary Sjögren's syndrome (SS) patients.

Currently, corticosteroids are the first-line therapy for CTD-associated thrombocytopenia, with second-line options including immunosuppressive agents, intravenous immunoglobulin (IVIG), splenectomy, and rituximab. However, not all patients respond favorably to these treatments. Patients with CTD who are unresponsive or have a low response to conventional first- and second-line therapies, with platelet counts below 30×10^9/L, are considered to have CTD-related refractory ITP (RITP). There are currently no internationally unified diagnostic criteria for RITP. For adult RITP diagnosis, criteria proposed by George et al. include: being diagnosed with ITP under the premise that treatment with glucocorticoids and/or splenectomy is ineffective; age ≥18 years; ③ duration of illness >6 months; ④ absence of other conditions causing thrombocytopenia; ⑤ platelet count ≤30×10^9/L.

Eltrombopag is an oral, small-molecule, non-peptide thrombopoietin receptor agonist that interacts with the transmembrane domain of the thrombopoietin receptor, stimulating platelet production and increasing platelet counts. To evaluate the efficacy and safety of eltrombopag in CTD-RITP, this study will conduct a single-center retrospective observational analysis of 52 patients with CTD-RITP who received eltrombopag treatment between 2013 and 2023, recording their follow-up information. Patient characteristics at baseline will be analyzed, and drug efficacy and safety will be assessed through follow-up examinations at different time points.

During treatment, patients may receive other ITP medications for maintenance therapy (such as glucocorticoids, azathioprine, danazol, cyclosporine A, and mycophenolate mofetil), excluding those concurrently using other TPO receptor agonists. Patient follow-up examinations will be continuously recorded (for at least six months, with monthly records, and patients followed until the last follow-up time if less than six months). Univariate analysis (descriptive analysis or non-parametric tests), single and multiple logistic regression analysis, and multiple correspondence analysis (MCA) will be used to analyze early clinical predictive factors for drug response. Patient drug responsiveness will be judged based on laboratory test results and clinical symptoms: ① Complete remission (CR): PLT ≥100×10^9/L with no bleeding tendency; ② Partial remission (PR): PLT ≥50×10^9/L but <100×10^9/L with no bleeding tendency, or platelet count at least twice that of pre-treatment; ③ No remission (NR): Does not meet criteria ① or ②. Mann-Kendall test will be used to analyze trends in PLT changes among patients during treatment, and the rates of CR, PR, and NR at different time points (4, 8, 12, 24 weeks) will be calculated to determine drug onset time and remission degree. The incidence of major adverse reactions to eltrombopag (hepatotoxicity, thrombosis) will be statistically analyzed at 24 weeks to assess drug safety.

This project aims to evaluate the efficacy and safety of eltrombopag in treating CTD-RITP patients, providing evidence for formulating treatment plans for CTD-RITP patients. It aims to guide physicians in considering the use of eltrombopag when selecting treatment methods, understanding individual differences in patient response to eltrombopag efficacy, and helping physicians develop more personalized treatment plans based on early clinical predictive factors to improve treatment targeting and effectiveness. Furthermore, it aims to observe the long-term effects of eltrombopag treatment and explore the optimal dosage, course of treatment, and best combination therapy with other drugs.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is diagnosed with CTD, SLE, SS, APS, MCTD, ANCA or RA according to international diagnostic criteria;
2. The patient meets the diagnostic criteria of RITP: (i) glucocorticoid therapy and/or splenectomy is ineffective; (ii) age ≥18 years; (iii) duration of the disease >6 months; (iv) no other diseases leading to thrombocytopenia; (v) platelet count ≤30×109/L;
3. At the time of enrolment, patients have received ineffective conventional first-line treatment for one year or more;
4. Enrolled patients need to be aware of the clinical information they are being given.

Exclusion Criteria:

1. The patient has a history of lymphoproliferative disease or malignancy of any organ system within the last 5 years;
2. The patient has a combination of other autoimmune diseases or malignant haematological diseases;
3. Patient's intermittent use of medication and failure to take medication as prescribed;
4. Patient refuses to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, a total of 52 CTD patients fulfilling refractory ITP criteria were enrolled, and all received oral eltrombopag at 25 to 75 mg once daily after failing to respond to conventional treatment of corticosteroids for more than one year. The time of follow-up ranged from 1 month to 15 months.
  1. Age at diagnosis, median (IQR) 45(34-60)
  2. Female, n (%) 43(82.7)
  3. SLE, n (%) 28(53.9)
  4. SS, n (%) 15(28.9)
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2013-05-06 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-11-19 (Actual)

PRIMARY OUTCOMES:
platelet counts of 52 patients from baseline after taking eltrombopag (Therapeutic effects-for refractory CTD-related ITP) | Baseline, post-intervention week 4, post-intervention week 8, post-intervention week 12, post-intervention week 24
  Platelet counts are measured to determine remission status (CTD-RITP). Partial remission is defined as platelet counts ≥ 50 × 10^9/L, and complete remission is defined as platelet counts ≥ 100 × 10^9/L.

SECONDARY OUTCOMES:
changes in disease activity index (Systemic Lupus Erythematosus Disease Activity Index 2000 for SLE patients and EULAR Sjögren's Syndrome Disease Activity Index 2000 for pSS patients) from baseline after taking Eltrombopag | Baseline, post-intervention week 4, post-intervention week 8, post-intervention week 12, post-intervention week 24
  Disease activities are measured in SLE patients by the SLEDAI (systemic lupus erythematosus disease activity index 2000) and in SS patients by the ESSDAI (EULAR Sjögren's syndrome disease activity index 2000), which indicate patients' remission from treatment. For Systemic Lupus Erythematosus Disease Activity Index 2000, the minimum score is 0 and the maximum score is 105. With a score of 5 or more, the disease is considered active. For EULAR Sjögren's Syndrome Disease Activity Index 2000, the minimum score is 0 and the maximum score is 51. With a score of 5 or more, the disease is considered active. The lower the disease activity, the more effective Eltrombopag is.

CONTACTS AND LOCATIONS:
Overall Officials: Lingli Dong, MD, Principal Investigator — Tongji Hospital

IPD SHARING:
Plan to Share IPD: Undecided